CLINICAL TRIAL: NCT01303614
Title: Lidocaine-Prilocaine (EMLA) Cream as Analgesia in Hysterosalpingography Practice: a Prospective Randomized Double Blind, Placebo-controlled Clinical Trial
Brief Title: Lidocaine-Prilocaine (EMLA) Cream as Analgesia in Hysterosalpingography Practice
Acronym: HSG-2010
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Consorci Sanitari de Terrassa (Other)
Responsible Party: Baldomero Arnau Rivera, Consorci Sanitari de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hysterosalpingography-2010
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2010-09

CONDITIONS: Gynecological Pathology
Keywords: hysterosalpingography; prilocaine; local anaesthetic; pain relief; gynecological pathology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine-Prilocaine cream (Active Comparator)
  Interventions: Drug: Lidocaine-Prilocaine cream
- Placebo (Placebo Comparator): purified water, ethylene glycol stearate, palm, palm stearate, polyethylene glycol, liquid paraffin, benzoic acid
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lidocaine-Prilocaine cream — Implementation of 3 cm of lidocaine-prilocaine in the endocervical canal, 10 minutes before the intervention with a syringe without needle 5ml. Application, with a swab of the anesthetic cream ectocervix level.
  Other Names: EMLA
  Arms: Lidocaine-Prilocaine cream
Drug: placebo — 3 cm of gel application for the transmission of ultrasound into the endocervical canal 10 minutes before surgery, with a 5 ml syringe without needle. Application, with a swab in gel ectocervix.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that Lidocaine-Prilocaine cream decrease pain during hysterosalpingography diagnostic practice.

ELIGIBILITY:
Inclusion Criteria:

* patients that must perform a hysterosalpingography
* acceptance to participate in the study signed informed consent

Exclusion Criteria:

* hypersensitivity or allergy to anesthetics
* refusal of the patient
* patients under age 18 years old and pregnant
* unbearable pain that involves other analgesic measures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
pain reduction in the performance of hysterosalpingography | after hysterosalpingography and a month later
  decrease in pain inmediately after the completion of hysterosalpingography and one month after completion of the diagnostic test by an analogue pain scale.

SECONDARY OUTCOMES:
sense of discomfort experience during the procedure | a month after hysterosalpingography
  willingness to repeat the diagnostic technique

CONTACTS AND LOCATIONS:
Overall Officials: Baldomero Arnau Rivera, MD, PhD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Derived] Arnau B, Jovell E, Romero M, Gonzalez M, Esteba L, Garcia A. Lidocaine-prilocaine cream as analgesia for hysterosalpingography: a randomized, double blinded, controlled study. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:216-9. doi: 10.1016/j.ejogrb.2014.09.035. Epub 2014 Sep 30. PMID 25445103